CLINICAL TRIAL: NCT05494775
Title: Effects of Corona Virus Pandemic on Intravitreal Injections
Brief Title: Effect of Corona Virus on Intravitreal Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Associate professor of Ophthalmology, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc-11-2022
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Macular Edema; Age-Related Macular Degeneration; Choroidal Neovascularization; Myopic Choroidal Neovascularisation; Diabetic Retinopathy
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diabetic macular edema (Active Comparator): Cases with diabetic macular edema that are prepared for intravitreal injection of anti-vascular endothelial growth factors.
  Interventions: Drug: Anti-vascular endothelial growth factors (Anti-VEGFs)
- Wet age related macular edema (Active Comparator): Cases with wet age related macular degenerations that are prepared for intravitreal injection of anti-vascular endothelial growth factors.
  Interventions: Drug: Anti-vascular endothelial growth factors (Anti-VEGFs)
- Retinal vein occlusion (Active Comparator): Cases with macular edema secondary to retinal vein occlusion that are prepared for intravitreal injection of anti-vascular endothelial growth factors.
  Interventions: Drug: Anti-vascular endothelial growth factors (Anti-VEGFs)
- Myopic choroidal new vascularization (Active Comparator): Cases with myopic choroidal new vascularization that are prepared for intravitreal injection of anti-vascular endothelial growth factors.
  Interventions: Drug: Anti-vascular endothelial growth factors (Anti-VEGFs)

INTERVENTIONS:
Drug: Anti-vascular endothelial growth factors (Anti-VEGFs) — Intravitreal injection of anti-vascular endothelial growth factors (Anti-VEGFs).

SUMMARY:
During pandemic of corona virus, patients compliance may be affected. We aim to study the factors lead to unregulated visits and its implications on the final visual outcome.

DETAILED DESCRIPTION:
The corona virus pandemic may affects patients regular visits to ophthalmic clinic, we aim to study the sequel of the pandemic on intravitreal injections results in diabetic macular edema, wet age related macular degenerations, myopic choroidal new vascularization, and proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with the following conditions (diabetic macular edema, wet age related macular degeneration, myopic choroidal new vascularization and retinal vein occlusion complicated with macular edema).

Exclusion Criteria:

* patients that are known to have hypersensitivity to Anti-VEGFs.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-06-11 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Baseline and monthly after injection till one year of follow-up
  Assessing the changes in best corrected visual acuity in logMAR unit measured by snellen chart.

SECONDARY OUTCOMES:
Central subfield thickness | Baseline and monthly after injection till one year of follow-up
  Assessing the changes in central macular thickness in microns measured by optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No